CLINICAL TRIAL: NCT05610787
Title: EXCOR Active Driving System for the EXCOR Pediatric VAD IDE Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Berlin Heart, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G200252
Record Dates: First submitted 2022-09-14; First posted 2022-11-09 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-12

CONDITIONS: Heart Failure; Transplant; Failure, Heart; Congenital Heart Disease
Keywords: Pediatric Ventricular Assist Device; Berlin Heart
MeSH Terms: conditions — Heart Failure; Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Open Label, Single Arm, Prospective, Non-Randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active Driver Primary Arm (Experimental): Up to 40 patients whom receive the Active Driver from implant.
  Interventions: Device: EXCOR Active Driving System for Pediatric VAD
- IKUS Comparator (No Intervention): All patients whom receive the (FDA approved) IKUS Driver from implant and are entered into the ACTION Registry.

INTERVENTIONS:
Device: EXCOR Active Driving System for Pediatric VAD — The EXCOR Active Driving System - will be used with the EXCOR Pediatric VAD.
  Arms: Active Driver Primary Arm

SUMMARY:
The purpose of this study is to evaluate the device performance and monitor the safety and effectiveness of the Berlin Heart EXCOR Active Driving System while being used with the approved EXCOR Pediatric Ventricular Assist Device.

EXCOR Active Driving System is intended for use with the approved EXCOR Pediatric VAD.

The EXCOR Pediatric VAD is intended to provide mechanical circulatory support as a bridge to cardiac transplantation for pediatric patients. Pediatric candidates with severe isolated left ventricular or biventricular dysfunction who are candidates for cardiac transplant and require circulatory support may be treated using the EXCOR Pediatric.

EXCOR Active is intended for use in a clinical setting. EXCOR Active can be used in any kind of hospital unit (e.g. OR, ICU, intermediate care unit or general care unit). The driving unit may be moved between clinical units using the caddy or baby buggy; however, a patient must always be accompanied by a person trained in the use of the manual pump and emergency procedures during transport in the event of an emergency.

The driving unit can be transported during operation.

DETAILED DESCRIPTION:
This is a prospective study of subjects implanted with the EXCOR Pediatric VAD supported by the EXCOR Active Driving System and patients recently implanted with EXCOR Pediatric supported on the Ikus Driving Unit as reported in the ACTION Registry database.

Children who are transplant eligible in need of mechanical circulatory support and are supported with the EXCOR® Pediatric VAD will be included in this study. All patients must meet the indications and contraindication as indicated in the device labelling. There are no known additional indications or contraindications associated with the EXCOR® Active Driving System beyond those already established in the EXCOR® Pediatric VAD labeling.

The objective of this study is to evaluate device performance and monitor safety and effectiveness of the Berlin Heart EXCOR® Active Driving System while being used with the approved EXCOR® Pediatric Ventricular Assist Device.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets all indications as specified in the current version of the Instructions for Use (IFU) of the EXCOR® Pediatric VAD system as shown below:

"EXCOR is intended to provide mechanical circulatory support as a bridge to cardiac transplantation for pediatric patients. Pediatric patients with severe isolated left ventricular or biventricular dysfunction who are candidates for cardiac transplant and require circulatory support may be treated using EXCOR."

• Patient and/or legal representative has signed the study informed consent form.

Exclusion Criteria:

• Patient has any contraindication as specified in the current version of the IFU of the EXCOR® Pediatric VAD system as shown below:

"Patients unable to tolerate systemic anticoagulation therapy should not be implanted with EXCOR components.

Magnetic Resonance Imaging (MRI) is contraindicated in patients after being implanted with EXCOR.

Patients with aortic valve regurgitation that is more than moderate that cannot be re- paired at the time of implantation should not be implanted with EXCOR. If repair of the aortic valve regurgitation requires surgical closure of the aortic valve, EXCOR should not be implanted. EXCOR is not intended to be used as a total artificial heart and should not be used in this configuration."

* Patient and/or legal representative has not given written consent to participate in the study (non-consent).
* Females of childbearing age who are not on contraceptives or surgically sterile or pregnant.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Device Malfunction adverse events | Up to 90 days
  A Device Malfunction per protocol definition, and adjudicated by the Clinical Events Committee.
Patient Outcome | Up to 90 days
  Patient outcomes will be summarized as the proportion of subjects experiencing each outcome and the overall successful outcome. Successful outcome is defined as:
  * survival to recovery/successful weaning -or-
  * survival to explantation not attributed to device malfunction -or-
  * survival on EXCOR® Pediatric at 90 days post-implant
  Patients who are removed from support followed by death or for escalation to other therapy (such as another VAD or ECMO) due to major device malfunction attributed to the Active Driving System will be considered failures.
Serious Adverse Events | Up to 90 days
  Serious Adverse Event rates will be calculated as the rate per 100 patient-months for each individual event as defined in protocol.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital-Stanford, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National, Washington D.C., District of Columbia
  - Boston Children's Hospital, Boston, Massachusetts
  - St Louis Children's Hospital, St Louis, Missouri
  - Levine Children's Hospital, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No